CLINICAL TRIAL: NCT06852846
Title: Clinical Usefulness of a Multi-analyte Immunoassay for Distinguishing Bacterial and Viral Infections in a Cohort of Pediatric Febrile Patients
Brief Title: Clinical Usefulness of a Multi-analyte Immunoassay for Distinguishing Bacterial and Viral Infections in Children
Acronym: PED_BIOMARKERS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Elisabetta Venturini, MD, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PED_BIOMARKER
Record Dates: First submitted 2025-02-20; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Febrile Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic Test (Other): Patients with fever (body temperature ≥38°C) for less than 7 days
  Interventions: Diagnostic Test: Biological sample

INTERVENTIONS:
Diagnostic Test: Biological sample — Biomarker test for tumor necrosis factor-related apoptosis-inducing ligand (TRAIL), interferon gamma-inducible protein of 10 kDa (IP-10), and C-reactive protein

SUMMARY:
Fever can be a clinical manifestation present in pediatric infections, posing a challenge for the doctor who must decide whether or not to prescribe an antibiotic therapy. Routine blood tests can assist the doctor in making a decision, although their response times often do not allow for timely therapeutic decisions. Therefore, there is an increased risk of inappropriate prescribing antibiotics for children with viral infections, which contributes to the increase in antibiotic resistance. There is evidence suggesting the effectiveness of certain biomarkers in distinguishing viral from bacterial forms. Biomarkers of potential interest include tumor necrosis factor-related apoptosis-inducing ligand (TRAIL), interferon gamma-inducible protein of 10 kDa (IP-10), and C-reactive protein. The combination of those tests could distinguish between bacterial and viral infections with 90-94% sensitivity, 88-92.8% specificity, 59-81% positive predictive value and 97-98.8% negative predictive value. This is prospective study using biological samples that aims to evaluate the best diagnostic algorithm for obtaining an early and accurate etiological diagnosis (bacterial infection vs viral infection) of a febrile pediatric patient presenting at the Emergency Department, by comparing the standard algorithm with the diagnostic algorithm integrated with the results of the multi-analytic test.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 3 months and < 18 years
* Access to the Emergency Department during the study period
* Fever (body temperature ≥38°C) for less than 7 days
* Absence of an infectious focus or symptoms affecting the respiratory tract

Exclusion criteria:

* Fever for more than 7 days
* Antibiotic therapy for ≥ 48 hours
* Acute gastroenteritis
* HBV (hepatitis B virus) or HCV (hepatitis C virus) infection
* Active oncologic pathology
* Metabolic pathology
* Trauma or major surgery within the past 7 days

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with concordance between biochemical test result and clinical diagnosis | From the date of enrollment to the date of diagnosis

CONTACTS AND LOCATIONS:
Locations (1):
- Meyer Children's Hospital IRCCS, Firenze, Florence, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papan C, Argentiero A, Adams O, Porwoll M, Hakim U, Farinelli E, Testa I, Pasticci MB, Mezzetti D, Perruccio K, Simon A, Liese JG, Knuf M, Stein M, Yacobov R, Bamberger E, Schneider S, Esposito S, Tenenbaum T. Association of viral load with TRAIL, IP-10, CRP biomarker signature and disease severity in children with respiratory tract infection or fever without source: A prospective, multicentre cohort study. J Med Virol. 2023 Jan;95(1):e28113. doi: 10.1002/jmv.28113. Epub 2022 Sep 9. PMID 36043485